CLINICAL TRIAL: NCT04336592
Title: Pilot Testing a Pain Management Intervention Preparatory to a Future Pragmatic Trial (NOHARM)
Brief Title: Pain Management Intervention Preparatory to a Future Pragmatic Trial
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jon C. Tilburt, Principal Investigator, Mayo Clinic
Other Study IDs: 20-001864; UG3AG067593 (NIH)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Non-Pharmacological Pain Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients scheduled to receive a surgical spine procedure at Mayo Clinic
  Interventions: Behavioral: Non-pharmacological Options in post-operative Hospital and Rehabilitative Management (NOHARM)
- Clinicians: Surgeons, Physician pain specialists and allied health caring for participating patients
  Interventions: Behavioral: Non-pharmacological Options in post-operative Hospital and Rehabilitative Management (NOHARM)

INTERVENTIONS:
Behavioral: Non-pharmacological Options in post-operative Hospital and Rehabilitative Management (NOHARM) — Gathers patient preferences for non-pharmacological pain management strategies through medical record and inform clinicians (via prompts, orders, etc.) of these preferences and encourages conversation about these preferences throughout their routine pre- and post-surgical interactions with patients. Resources will be provided to bedside clinicians as they assist patients in identifying a personalized post-discharge pain management strategy.

SUMMARY:
Researchers are promoting non-pharmacological pain management strategies for patients by assisting them in identifying post-surgical pain care preference following an operative procedure at Mayo Clinic.

DETAILED DESCRIPTION:
This is a pilot study to test promoting non-pharmacological pain management strategies for patients by assisting them in identifying post-surgical pain care preference following an operative procedure. This pilot study will confirm the feasibility of patient-facing as well as clinician-facing decision support components of an electronic health record (EHR) imbedded evidence-based bundle.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to receive a surgical spine procedure at Mayo Clinic
* Surgeons, Physician pain specialists and allied health caring for patients meeting patient inclusion criteria

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to receive a surgical procedure at Mayo Clinic and their clinicians involved in the care.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Non-Pharmacological options participation | 1 month post-operative
  Number of participants to complete the non-pharmacological options in post-operative Hospital and Rehabilitative Management

CONTACTS AND LOCATIONS:
Overall Officials: Jon Tilburt, MD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System - Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic Health System - Franciscan Healthcare, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials